CLINICAL TRIAL: NCT00993161
Title: Development and Evaluation of a Clinical Test in Order Quantify Muscular Function in Upper Limb of Non Ambulatory Patients With Neuromuscular Disorder
Brief Title: Upper Limb Evaluation in Non Ambulatory Patients With Neuromuscular Disorder
Acronym: ULENAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ULENAP
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Neuromuscular Disorders
Keywords: Neuromuscular disorders; Evaluation; Strength; Upper limb
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Experimental): Patients with neuromuscular disorder and controls
  Interventions: Device: Motriplate
- Controls (Experimental): healthy controls
  Interventions: Device: Motriplate

INTERVENTIONS:
Device: Motriplate — Number of contact couples
  Arms: patients
Device: Motriplate — Number of contact couples
  Arms: Controls

SUMMARY:
The aim of this study is to evaluate different devices to quantify upper limb function (Motriplate) and strength (Myogrip, Myopinch) in non-ambulatory patients with neuromuscular disorder. Motriplate measures the ability of the patient to reproduce a repetitive movement of the wrist to push two 5cm*5cm targets during 30 seconds. One hundred patients aged 8-30 years and 60 controls will be evaluated during twelve months (M0, M6 and M12) with theses new tools, and results will be compared to other testing, such as wrist, grip and pinch strength, taping, MFM measurement, and self evaluation of hand ability.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed neuromuscular disorder
* Aged 8-30 years
* Written consent
* Non ambulant

Exclusion Criteria

* Major cognitive impairment
* Inability to stay seated one hour
* Recent upper limb surgery or trauma
* Treatment by steroids initiated less than 6 months before

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 174 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of contact couples with the targets | Month 0, Day 60, Month 6, Month 12

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Raymond Poincare, Garches
  - Trousseau, Paris
  - Institut de Myologie, Paris
  - Necker, Paris

REFERENCES:
- [Background] Mercuri E, Mayhew A, Muntoni F, Messina S, Straub V, Van Ommen GJ, Voit T, Bertini E, Bushby K; TREAT-NMD Neuromuscular Network. Towards harmonisation of outcome measures for DMD and SMA within TREAT-NMD; report of three expert workshops: TREAT-NMD/ENMC workshop on outcome measures, 12th--13th May 2007, Naarden, The Netherlands; TREAT-NMD workshop on outcome measures in experimental trials for DMD, 30th June--1st July 2007, Naarden, The Netherlands; conjoint Institute of Myology TREAT-NMD meeting on physical activity monitoring in neuromuscular disorders, 11th July 2007, Paris, France. Neuromuscul Disord. 2008 Nov;18(11):894-903. doi: 10.1016/j.nmd.2008.07.003. Epub 2008 Sep 24. No abstract available. PMID 18818076
- [Derived] Seferian AM, Moraux A, Canal A, Decostre V, Diebate O, Le Moing AG, Gidaro T, Deconinck N, Van Parys F, Vereecke W, Wittevrongel S, Annoussamy M, Mayer M, Maincent K, Cuisset JM, Tiffreau V, Denis S, Jousten V, Quijano-Roy S, Voit T, Hogrel JY, Servais L. Upper limb evaluation and one-year follow up of non-ambulant patients with spinal muscular atrophy: an observational multicenter trial. PLoS One. 2015 Apr 10;10(4):e0121799. doi: 10.1371/journal.pone.0121799. eCollection 2015. PMID 25861036
- [Derived] Seferian AM, Moraux A, Annoussamy M, Canal A, Decostre V, Diebate O, Le Moing AG, Gidaro T, Deconinck N, Van Parys F, Vereecke W, Wittevrongel S, Mayer M, Maincent K, Desguerre I, Themar-Noel C, Cuisset JM, Tiffreau V, Denis S, Jousten V, Quijano-Roy S, Voit T, Hogrel JY, Servais L. Upper limb strength and function changes during a one-year follow-up in non-ambulant patients with Duchenne Muscular Dystrophy: an observational multicenter trial. PLoS One. 2015 Feb 2;10(2):e0113999. doi: 10.1371/journal.pone.0113999. eCollection 2015. PMID 25643053
- See also: website of the sponsor — http://www.institut-myologie.org